CLINICAL TRIAL: NCT01602432
Title: Implementing a Tool to Identify Risk for Venous Thromboembolism in Cancer Patients
Status: Withdrawn | Type: Observational
Why Stopped: Project did not meet criteria of a research study and was confirmed as a Quality Initiative Project
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Other Study IDs: 20120209-01H
Record Dates: First submitted 2012-05-16; First posted 2012-05-21 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2014-09

CONDITIONS: Venous Thromboembolism; Deep-Vein Thrombosis; Pulmonary Embolism; Cancer
Keywords: Venous Thrombosis; Cancer; Coagulation factors; Blood
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High Risk Group: Defined as patients whose primary malignancy is located in the brain, bladder, lung, testicle, stomach, pancreas and lymphatic system and whose risk score before the beginning of anticancer treatment is ≥ 2 according to the Risk Stratification Method proposed by Khorana et al. (2008).
  Based on this method, the model includes 5 predictive variables as follows:
  1. Site of cancer: classified as very high-risk (+2 points) or high-risk (+1 point).
  2. Platelet count: (>350 x 109/L) (+1 point)
  3. Hemoglobin level (<100 g/L) and/or use of erythropoiesis stimulating agents (+1 point)
  4. Leukocyte count (> 11 x 109/L)(+1 point).
  5. body mass index (≥ 35 Kg/m2) (+1 point).
- Low high Risk Group: Defined as patients whose primary malignancy is located in the brain, bladder, lung, testicle, stomach, pancreas and lymphatic system and whose risk score before the beginning of anticancer treatment is < 2 according to the Risk Stratification Method proposed by Khorana et al. (2008).
  In order to confirm the patient low risk status, we will draw a blood sample to determine serum levels of D- dimer and soluble P selectin in patients of this low risk group according to Ay et al. (2010). If levels of D-dimer are ≥ 1.44 µg/mL and/or soluble P selectin ≥ 53.1 ng/mL, we will add one point for each one of the increased biochemical marker and the total score recalculated.

SUMMARY:
Cancer increases the risk of deep vein blood clots and clots traveling to the lungs (emboli) which cause morbidity (leg swelling, pain, and shortness of breath), sudden death, delays cancer treatment, and decreases cancer survival by 66% compared to similar cancer patients without blood clots. Blood thinners may prevent clots but major bleeding is also a problem, so preventive therapies are not used routinely. Identifying patients at highest risk for clots is critical. A tool exists but it has not been used outside of research. We propose to study how to apply this tool in clinical practice and test if it works.

DETAILED DESCRIPTION:
Patients with Cancer have a risk for venous thromboembolism (VTE) including deep-vein thrombosis (DVT) and/or pulmonary embolism (PE) that is markedly higher than non-Cancer patients. An acute episode of VTE has deleterious effects on the quality of life and long-term survival of cancer patients. Cancer patients with VTE have survival rates that are only one third of otherwise identical patients without VTE. Once VTE is diagnosed over 10% of cancer patients suffer a further event while on standard therapy and over 5% suffer a major hemorrhagic event.

The best way to treat VTE is its prevention (thromboprophylaxis). Studies suggest that among ambulatory cancer patients, risk for VTE varies markedly between patients and that the lack of knowledge of this risk, delays diagnosis and hampers efforts to effectively prevent VTE. Therefore, the identification of patients at high-risk for VTE may enable faster diagnosis of VTE and better use of thromboprophylaxis.

Recent studies have developed a novel tool to stratify VTE risk in cancer patients before they initiate anti-cancer treatment. We hypothesized that this risk tool will accurately identify cancer patients at high-risk and that its implementation in our clinical practice will result in a faster clinical diagnosis of VTE.

Our objective is: a) to evaluate the ideal strategy to incorporate the tool in our clinical setting as seamlessly as possible, and b) to determine whether the tool accurately predicts risk and results in a faster investigation for VTE.

Patient eligibility will be determined during the patient's initial consult to the Ottawa Cancer Center after cancer diagnosis has been confirmed by the medical Oncologist and before initiation of anticancer treatment. Follow-up for this study will be for 12 months and patients will be seen at the time of scheduled appointments for cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* with a newly diagnosed cancer site (brain, bladder, lung, testicle, pancreas, stomach and lymphomas)
* or progression of the malignant disease after complete or partial remission who have not recently received chemotherapy (≤ 3 months), radiotherapy and surgery (≤ 2 weeks)

Exclusion Criteria:

* Cancer patients with confirmed VTE or arterial embolism within the last 3 months
* Cancer patients who are receiving continuous anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Because of their higher thrombogenic potential, we will aim to identify high-risk cases for VTE within the group of cancer patients whose primary malignancy is located in the brain, bladder, lung, testicle, pancreas, stomach and lymphomas.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Risk for Venous Thromboembolism | 1 year
  This outcome will be measured by the cummulative rates of VTE stratified by the different categories of risk as determined by the prediction tool during the time-frame of the study

SECONDARY OUTCOMES:
Timing to VTE detection | 1 year
  This will be measured by the time elapsed between the first signs or symptoms associated with a symptomatic VTE as described by the patient and the time of confirming VTE diagnosis.
Study Feasibility | 1 year
  Feasibility will be assessed by: a) achieving an average enrollment rate of at least 39 cancer patients per month; and b) accomplishing a rate of withdrawals or loss to follow-ups equal or less than 10%
Physicians acceptance | 1 year
  This will be assessed by measurements of physician's satisfaction to the implementation of the Risk stratification tool at the end of the study period.
Success of an IS/IT solution | 1 year
  This outcome will be measured by the physician's satisfaction to the implementation of an automatic risk detection.

CONTACTS AND LOCATIONS:
Overall Officials: Philip S Wells, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Cancer Center, Ottawa, Ontario, Canada

REFERENCES:
- [Background] Noble S, Pasi J. Epidemiology and pathophysiology of cancer-associated thrombosis. Br J Cancer. 2010 Apr 13;102 Suppl 1(Suppl 1):S2-9. doi: 10.1038/sj.bjc.6605599. PMID 20386546
- [Background] Louzada ML, Majeed H, Dao V, Wells PS. Risk of recurrent venous thromboembolism according to malignancy characteristics in patients with cancer-associated thrombosis: a systematic review of observational and intervention studies. Blood Coagul Fibrinolysis. 2011 Mar;22(2):86-91. doi: 10.1097/MBC.0b013e328341f030. PMID 21245746
- [Background] Lee AY, Levine MN, Baker RI, Bowden C, Kakkar AK, Prins M, Rickles FR, Julian JA, Haley S, Kovacs MJ, Gent M; Randomized Comparison of Low-Molecular-Weight Heparin versus Oral Anticoagulant Therapy for the Prevention of Recurrent Venous Thromboembolism in Patients with Cancer (CLOT) Investigators. Low-molecular-weight heparin versus a coumarin for the prevention of recurrent venous thromboembolism in patients with cancer. N Engl J Med. 2003 Jul 10;349(2):146-53. doi: 10.1056/NEJMoa025313. PMID 12853587
- [Background] Khorana AA, Francis CW, Culakova E, Fisher RI, Kuderer NM, Lyman GH. Thromboembolism in hospitalized neutropenic cancer patients. J Clin Oncol. 2006 Jan 20;24(3):484-90. doi: 10.1200/JCO.2005.03.8877. PMID 16421425
- [Background] Khorana AA, Connolly GC. Assessing risk of venous thromboembolism in the patient with cancer. J Clin Oncol. 2009 Oct 10;27(29):4839-47. doi: 10.1200/JCO.2009.22.3271. Epub 2009 Aug 31. PMID 19720906
- [Background] Khorana AA, Kuderer NM, Culakova E, Lyman GH, Francis CW. Development and validation of a predictive model for chemotherapy-associated thrombosis. Blood. 2008 May 15;111(10):4902-7. doi: 10.1182/blood-2007-10-116327. Epub 2008 Jan 23. PMID 18216292
- [Background] Ay C, Dunkler D, Marosi C, Chiriac AL, Vormittag R, Simanek R, Quehenberger P, Zielinski C, Pabinger I. Prediction of venous thromboembolism in cancer patients. Blood. 2010 Dec 9;116(24):5377-82. doi: 10.1182/blood-2010-02-270116. Epub 2010 Sep 9. PMID 20829374
- [Background] Carrier M, Tay J, Fergusson D, Wells PS. Thromboprophylaxis for catheter-related thrombosis in patients with cancer: a systematic review of the randomized, controlled trials. J Thromb Haemost. 2007 Dec;5(12):2552-4. doi: 10.1111/j.1538-7836.2007.02751.x. No abstract available. PMID 18034768
- [Background] Stanley A, Young A. Primary prevention of venous thromboembolism in medical and surgical oncology patients. Br J Cancer. 2010 Apr 13;102 Suppl 1(Suppl 1):S10-6. doi: 10.1038/sj.bjc.6605600. PMID 20386544